CLINICAL TRIAL: NCT06363188
Title: The Impact of Using Extracorporeal Radial Shock Wave Therapy as an Adjuvant Therapy vs Conventional Open Reduction and Internal Fixation With No Adjuvant Therapy on Bone Healing for Patients With Mandibular Parasymphyseal, Body and Angle Fractures
Brief Title: The Impact of ESWT on Healing of Fractured Mandible
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khloud Ahmed Mohamed, Khloud Ahmed Mohamed Hussien, Cairo University
Other Study IDs: effect of ESWT on fractures
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Fractured Mandible Due to Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- intervention group: Firstly the patient is generally anesthetized by the anesthesiologist. Intermaxillary fixation (IMF) screws has been inserted in case of there is no arch bar is used.
  The transoral or extraoral approach is utilized to expose the fracture line separating the two segments.
  Fixation of the bony segments with two plates one Compression 2.3 plate at the inferior border and Tension 2.0 plate five millimeter superiorly to the compression plate.
  or 1 plate2.0 (champy) Then suturing the incision layers Postoperative evaluation with cone beam computed tomography (CBCT). These procedures will be done for both groups. This group will be subjected to shockwave by the usage of extracorporeal shockwave device at the third day postoperative.
  Then follow up at the first and fourth month with another CBCT to compare the bone healing at the fracture site.
  Interventions: Device: Radial Extracorporeal shockwave
- control group: Firstly the patient is generally anesthetized by the anesthesiologist. Intermaxillary fixation (IMF) screws has been inserted in case of there is no arch bar is used.
  The transoral or extraoral approach is utilized to expose the fracture line separating the two segments.
  Fixation of the bony segments with two plates one Compression 2.3 plate at the inferior border and Tension 2.0 plate five millimeter superiorly to the compression plate.
  or 1 plate2.0 (champy) Then suturing the incision layers Postoperative evaluation with cone beam computed tomography (CBCT). The control group with no adjuvant intervention will stop at this point. Then follow up at the first and fourth month with another CBCT to compare the bone healing at the fracture site.

INTERVENTIONS:
Device: Radial Extracorporeal shockwave — a device used by physiotherapist to treat various musculoskeletal problems and it was here firstly used to accelerate the bone healing process after bone fracture
  Groups: intervention group

SUMMARY:
studying if using extracorporeal radial shockwave therapy as an adjuvant therapy help in accelerating the bone healing and regeneration in mandibular fractures by comparing it with the standard protocol for fractures fixation by plates and screws.

DETAILED DESCRIPTION:
Firstly the patient heads to the operating room being placed in a supine position, generally anesthetized by the anesthesiologist.

Sterilization of intraoral and extraoral sites and draping has been installed. Intermaxillary fixation (IMF) screws has been inserted in case of there is no arch bar is used.

If the arch bar has been used it was inserted before the operation and being cut at the fracture line between the two segments.

The transoral or extra-oral approach is utilized to expose the fracture line separating the two segments.

Fixation of the bony segments with two plates one Compression 2.3 plate at the inferior border and Tension 2.0 plate five millimeter superiorly to the compression plate.

or even one 2.0 plate(champy) Then suturing the incision layers with vicryl 3/0. Postoperative evaluation with cone beam computed tomography (CBCT). These procedures will be done for both groups. The control group with no adjuvant intervention will stop at this point. The other intervention group will be subjected to shockwave by the usage of extracorporeal shockwave device at the third day postoperative.

Then follow up at the first and fourth month with another CBCT to compare the bone healing at the fracture site.

ELIGIBILITY:
Inclusion Criteria:

1 - Patients with age ranges from 18-75 years old. 2- Patients with fresh mandibular fractures (from zero hour till four or five days).

3- Patients free of systemic conditions that might affect or interfere with the healing process of bone segments or rather interfere with carrying out the surgical procedure (thyroid condition, rheumatoid arthritis, uncontrolled diabetes and osteoporosis).

Exclusion Criteria:

1 - Patients out of the specified range group 2- Patients who went previous operations with infection or malunion. 3- Patients with thyroid condition which affects the serum calcium level. 4- Patients with systemic conditions that might affect the bone health (osteoarthritis, rheumatoid arthritis, uncontrolled diabetes). 5- Patients with heart peacemakers.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Patients with age ranges from 18-75 years old.
  2. Patients with fresh mandibular fractures (from zero hour till four or five days).
  3. Patients free of systemic conditions that might affect or interfere with the healing process of bone segments or rather interfere with carrying out the surgical procedure (thyroid condition, rheumatoid arthritis, uncontrolled diabetes and osteoporosis).
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
bone healing (denisty of bone) | first and fourth month
  radiographically we will analyze the bone denisty at the fracture site

SECONDARY OUTCOMES:
pain sensation | immediately after the intervention and 3 days after
  depending on the patient using VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Univeristy, Cairo, Egypt

REFERENCES:
- [Background] Verma S, Chambers I. Update on patterns of mandibular fracture in Tasmania, Australia. Br J Oral Maxillofac Surg. 2015 Jan;53(1):74-7. doi: 10.1016/j.bjoms.2014.10.003. Epub 2014 Nov 1. PMID 25453253
- [Background] Sirimaharaj W, Pyungtanasup K. The epidemiology of mandibular fractures treated at Chiang Mai University Hospital: a review of 198 cases. J Med Assoc Thai. 2008 Jun;91(6):868-74. PMID 18697387
- [Background] Chocron Y, Azzi AJ, Davison P. Management of Pediatric Mandibular Fractures Using Resorbable Plates. J Craniofac Surg. 2019 Oct;30(7):2111-2114. doi: 10.1097/SCS.0000000000006002. PMID 31568159
- [Background] Fridrich KL, Pena-Velasco G, Olson RA. Changing trends with mandibular fractures: a review of 1,067 cases. J Oral Maxillofac Surg. 1992 Jun;50(6):586-9. doi: 10.1016/0278-2391(92)90438-6. PMID 1593318
- [Background] Lamphier J, Ziccardi V, Ruvo A, Janel M. Complications of mandibular fractures in an urban teaching center. J Oral Maxillofac Surg. 2003 Jul;61(7):745-9; discussion 749-50. doi: 10.1016/s0278-2391(03)00147-2. PMID 12856243
- [Background] Ellis E 3rd. Complications of rigid internal fixation for mandibular fractures. J Craniomaxillofac Trauma. 1996 Summer;2(2):32-9. PMID 11951481
- [Background] Cacchio A, Giordano L, Colafarina O, Rompe JD, Tavernese E, Ioppolo F, Flamini S, Spacca G, Santilli V. Extracorporeal shock-wave therapy compared with surgery for hypertrophic long-bone nonunions. J Bone Joint Surg Am. 2009 Nov;91(11):2589-97. doi: 10.2106/JBJS.H.00841. PMID 19884432
- [Background] Kaspar D, Neidlinger-Wilke C, Holbein O, Claes L, Ignatius A. Mitogens are increased in the systemic circulation during bone callus healing. J Orthop Res. 2003 Mar;21(2):320-5. doi: 10.1016/S0736-0266(02)00134-1. PMID 12568965
- [Background] Heller GZ, Manuguerra M, Chow R. How to analyze the Visual Analogue Scale: Myths, truths and clinical relevance. Scand J Pain. 2016 Oct;13:67-75. doi: 10.1016/j.sjpain.2016.06.012. Epub 2016 Jul 27. PMID 28850536